CLINICAL TRIAL: NCT01259804
Title: Efficacy and Safety of High-dose Peanut Oral Immunotherapy With Factors Predicting Outcome
Brief Title: Study of Tolerance to Oral Peanut
Acronym: STOP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dr. Andrew Clark, Consultant, Cambridge University Hospitals NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STOP-I
Record Dates: First submitted 2010-12-13; First posted 2010-12-14 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Peanut Allergy
Keywords: peanut; food allergy; anaphylaxis; immunotherapy
MeSH Terms: conditions — Peanut Hypersensitivity; Food Hypersensitivity; Anaphylaxis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Peanut immunotherapy (Experimental): Peanut flour
  Interventions: Dietary Supplement: Peanut oral immunotherapy

INTERVENTIONS:
Dietary Supplement: Peanut oral immunotherapy — Daily doses of peanut flour
  Other Names: Daily doses peanut flour

SUMMARY:
Open pilot study of peanut oral immunotherapy in 22 children with peanut allergy

DETAILED DESCRIPTION:
Background Peanut allergy is severe and rarely resolves.

Objective To test the efficacy and safety of a new oral immunotherapy protocol for peanut allergy.

Method 22 peanut-allergic children will undergo oral challenge. Oral immunotherapy will be administered by gradual updosing with 2-weekly increments (8-38w) to 800mg protein (5 peanuts/day) followed by 30-weeks maintenance. Oral challenge will be repeated after 6 and 30 weeks maintenance.

ELIGIBILITY:
Inclusion Criteria:

* Peanut allergy defined by oral challenge

Exclusion Criteria:

* Major immunodeficiency

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2008-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Pass/fail peanut challenge | six months

CONTACTS AND LOCATIONS:
Overall Officials: Andrew T Clark, MB BD MD, Principal Investigator — Cambridge Biomedical Campus
Locations (1):
- Cambridge Biomedical Campus, Cambridge, Cambridgeshire, United Kingdom

REFERENCES:
- [Result] Clark AT, Islam S, King Y, Deighton J, Anagnostou K, Ewan PW. Successful oral tolerance induction in severe peanut allergy. Allergy. 2009 Aug;64(8):1218-20. doi: 10.1111/j.1398-9995.2009.01982.x. Epub 2009 Feb 17. PMID 19226304
- [Derived] Santos AF, James LK, Kwok M, McKendry RT, Anagnostou K, Clark AT, Lack G. Peanut oral immunotherapy induces blocking antibodies but does not change the functional characteristics of peanut-specific IgE. J Allergy Clin Immunol. 2020 Jan;145(1):440-443.e5. doi: 10.1016/j.jaci.2019.09.005. Epub 2019 Oct 30. No abstract available. PMID 31676085
- [Derived] Anagnostou K, Clark A, King Y, Islam S, Deighton J, Ewan P. Efficacy and safety of high-dose peanut oral immunotherapy with factors predicting outcome. Clin Exp Allergy. 2011 Sep;41(9):1273-81. doi: 10.1111/j.1365-2222.2011.03699.x. Epub 2011 Mar 18. PMID 21414048